CLINICAL TRIAL: NCT01250392
Title: The Effect of Time-Slot Scheduling and Active Choice on Biometric Screening and Nurse Visit Participation
Brief Title: The Effect of Active Choice on Nurse Visit Participation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Bureau of Economic Research, Inc. (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 0001; P30AG034532 (NIH)
Record Dates: First submitted 2010-11-29; First posted 2010-11-30 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Participation in Nurse Visits
Keywords: Active choice; Nurse visits; Behavioral economics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Arm (Other): The control group will be informed via e-mail of the window of dates during which they can take part in the on-site screening and given instructions for scheduling an appointment.
  Interventions: Behavioral: The Effect of Active Choice on Nurse Visit Participation
- Active Choice Only Arm (Experimental): The active choice only arm, will be given the same information as the control group, but they will also be asked to make an appointment immediately, defer the scheduling decision, or decline to receive a screening.
  Interventions: Behavioral: The Effect of Active Choice on Nurse Visit Participation

INTERVENTIONS:
Behavioral: The Effect of Active Choice on Nurse Visit Participation — The goal of this project is to see if active choice will increase an individual's likelihood of participating in a nurse visit.
  The employees in our sample will schedule their nurse visit time slot via e-mail and a health service provider website. The control group will be informed via e-mail of the window of dates during which they can take part in the on-site screening and given instructions for scheduling an appointment. The treatment group, the active choice only arm, will be given the same information as the control group, but they will also be asked to make an appointment immediately, defer the scheduling decision, or decline to receive a screening. The treatment group will also receive email reminders one week before their appointment.
  Other Names: Active Choice and Participation

SUMMARY:
The goal of this project is to see if behavioral nudges will increase an individual's likelihood of participating in a nurse visit. The behavioral nudges under consideration are encouraging subjects to make an active choice and sending reminders.

DETAILED DESCRIPTION:
The employees in our sample will schedule their nurse visit time slot via e-mail and a health service provider website. Much as is the case in the current system, the control group will be informed via e-mail of the window of dates during which they can take part in the on-site screening and given instructions for scheduling an appointment. The treatment group, the active choice only arm, will be given the same information as the control group, but they will also be asked to make an appointment immediately, defer the scheduling decision, or decline to receive a screening. The treatment group will also receive email reminders one week before their appointment.

ELIGIBILITY:
Inclusion Criteria:

* Harrah's employee
* Registered e-mail address with Harrah's
* Part of Harrah's Choosing Wellness Program

Exclusion Criteria:

* Under 18
* Already participated in a nurse visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3500 (Actual)
Dates: Start 2010-12; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Nurse Visit Participation | This will be measured after all of the nurse visit windows have been closed, by 4/30/11
  We will measure whether or not subjects scheduled and participated in a nurse visit. We will compare the number of subjects who participated in the nurse visits by treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: David I Laibson, Ph.D, Principal Investigator — National Bureau of Economic Research
Locations (1):
- Caesars Corporate Office, Las Vegas, Nevada, United States